CLINICAL TRIAL: NCT00986284
Title: Phase II Study of EGFR Status Based Gefitinib Neoadjuvant Therapy in NSCLC Patients
Brief Title: Epidermal Growth Factor Receptor (EGFR) Status Based Gefitinib Neoadjuvant Therapy in Non Small Cell Lung Cancer (NSCLC)
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of patients and some progressed disease soon after surgery
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TMU-CIH-LCC-001
Record Dates: First submitted 2009-09-27; First posted 2009-09-29 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2012-08

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Non Small Cell Lung Cancer; Gefitinib; Neoadjuvant Therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gefitinib, Neoadjuvant therapy (Experimental): Patients with EGFR mutation will be recruited and treated with gefitinib.
  Interventions: Drug: gefitinib

INTERVENTIONS:
Drug: gefitinib — Patients with EGFR mutation in exon 19 or 21 will be administrated with gefitinib as neoadjuvant therapy. Then evaluated for response and then operation for operable patients.
  Other Names: Iressa

SUMMARY:
This study aims to investigate the efficacy and safety of gefitinib as neoadjuvant therapy in stage IIIA NSCLC patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients pathological diagnosed with NSCLC,with EGFR sensitive mutation;
* Stage IIIA patients with technical operable disease evaluated by image and lab results;
* Patients without chemotherapy or targeted-therapy before;
* Inform Consent.

Exclusion Criteria:

* Patients with malignant tumor other than lung cancer;
* Patients with other diseases such as cardiovascular disease that may hamper follow up;
* Patients that may not coordinate well,judged by researcher.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2009-09; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Response Rate | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Changli Wang, MD, Study Director — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Cancer Institute & Hospital, Tianjin, Tianjin Municipality, China